CLINICAL TRIAL: NCT05700084
Title: Phase I Clinical Trial on Tolerability and Bioavailability of Utidelone Capsule in Patients With Advanced Solid Tumors
Brief Title: Tolerability and Bioavailability of Utidelone Capsule in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2101
Record Dates: First submitted 2022-12-30; First posted 2023-01-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor
Keywords: Tolerability; Bioavailability; Advanced Solid Tumor
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Study design: Part 1 is a dose-escalation trial, and it's an open design; Part 2 is for pharmacokinetic comparison and food effect study, and it's an open, controlled design. Part 3 is expansion test of utidelone capsule combined with capecitabine.
  In the Part 1 dose-escalation trial, there is no control; in the Part 2 pharmacokinetic comparison and food effect study, utidelone injection is chosen as the control drug in Cycle 0 and 1; in Cycle 2 day1, high-fat postprandial dosing is served as the control.Part 3: expansion test of utidelone capsule combined with capecitabine dosage administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Utidelone Capsule (Part 1) (Experimental): Utidelone Capsule, available as 10 mg/capsule and 15 mg /capsule. Doses between 50 mg/m2/d and 120 mg/m2/d administered orally will be explored. Patients will be dosed for 5/7 consecutive days in a 21 day cycle.
  Interventions: Drug: Utidelone Capsule (Part 1)
- Utidelone Capsule/Utidelone Injection (Group A-B, Part 2) (Experimental): At cycle 0, patients will take Utidelone Capsule in fasted status at 60 mg/m2/d. At cycle 1, patients will be administered Utidelone Injection by iv drip at 30 mg/m2/d. At Cycle 2, patients will take Utidelone Capsule (after meals) at 60 mg/m2/d.
  Interventions: Drug: Drug A Utidelone Capsule (Part 2: Group A-B); Drug: Drug B Utidelone Injection (Part 2: Group A-B)
- Utidelone Injection/Utidelone Capsule (Group B-A, Part 2) (Experimental): At cycle 0, patients will be administered Utidelone Injection by iv drip at 30 mg/m2/d. At cycle 1, patients will take Utidelone Capsule in fasted status at 60 mg/m2/d. At cycle 2, patients will take Utidelone Capsule (after meals) at 60 mg/m2/d.
  Interventions: Drug: Drug A Utidelone Capsule (Part 2: Group B-A); Drug: Drug B Utidelone Injection (Part 2: Group B-A)
- Utidelone Capsule combination with Capecitabine (Experimental): Dosage:
  Utidelone capsule: 60 mg/m2/d, administered once a day on an empty stomach, continuously for 5 days from day 1 to day 5, with a treatment cycle of 21 days.
  Capecitabine: 1000mg/m2, twice a day (daily dose 2000mg/m2), once in the morning and once in the evening, taken orally within 30 minutes after meals. It is administered continuously for 14 days from day 1 to day 14, with a 21 day treatment cycle.
  Interventions: Drug: Capecitabine; Drug: Utidelone Capsule (Part 3)

INTERVENTIONS:
Drug: Utidelone Capsule (Part 1) — At least 3 dose cohorts are planned, and 14-26 cases are expected. Cohort 1: 2 cases are planned, and the subjects will receive Utidelone Capsule at a dose of 50 mg/m2/d for 5 days.
  Other dose-escalation cohorts: 3-6 cases are planned in each cohort, following the 3 + 3 design. The subjects in these cohorts will receive Utidelone Capsule at 75 mg/m2/d for 5 days, 100 mg/m2/d for 5 days, 100 mg/m2/d for 7 days, and 120 mg/m2/d for 7 days, in a 21-day cycle respectively.
  Arms: Utidelone Capsule (Part 1)
Drug: Drug A Utidelone Capsule (Part 2: Group A-B) — Utidelone Capsule at Part 2 in Group A-B will be administered at 60 mg/m2/d.
  At Cycle 0, on day 1, all patients will receive the drug in fasted status with a glass (approximately 240 ml) of warm water (2 h of fasting before administration; 2 h of fasting after administration).
  At Cycle 2, subjects will receive the drug after meals on days 1-5 (high-fat meal, drug taken 30 min after the meal; 2 h fasting after administration). Subjects will receive the drug on day 1-5 with 21 days as a cycle.
  For the subsequent treatment period, there is no special requirements for food. Subjects will receive the drug on day 1-5 with 21 days as a cycle.
  Arms: Utidelone Capsule/Utidelone Injection (Group A-B, Part 2)
Drug: Drug A Utidelone Capsule (Part 2: Group B-A) — Utidelone Capsule at Part 2 in Group B-A will be administered at 60 mg/m2/d.
  At Cycle 1, on day 1-5, all patients will receive the drug in fasted status with a glass (approximately 240 ml) of warm water (2 h of fasting before administration; 2 h of fasting after administration), with 21 days as a cycle.
  At Cycle 2, subjects will receive the drug after meals on days 1-5 (high-fat meal, drug taken 30 min after the meal; 2 h fasting after administration), with 21 days as a cycle.
  For the subsequent treatment period, there is no special requirements for food. Subjects will receive the drug on day 1-5 with 21 days as a cycle.
  Arms: Utidelone Injection/Utidelone Capsule (Group B-A, Part 2)
Drug: Drug B Utidelone Injection (Part 2: Group A-B) — Utidelone Injection at Part 2 in Group A-B will be administered at 30 mg/m2/d in 250 mL normal saline, intravenous drip over1.5 h.
  For Cycle 1, subjects will be administered Utidelone Injection on day 1-5 with 21 days as a cycle.
  Arms: Utidelone Capsule/Utidelone Injection (Group A-B, Part 2)
Drug: Drug B Utidelone Injection (Part 2: Group B-A) — Utidelone Injection at Part 2 in Group B-A will be administered at 30 mg/m2/d in 250 mL normal saline, intravenous drip over1.5 h.
  For Cycle 0, all patients will be administered Utidelone Injection on day 1, with 21 days as a cycle.
  Arms: Utidelone Injection/Utidelone Capsule (Group B-A, Part 2)
Drug: Capecitabine — 1000mg/m2, twice a day (daily dose 2000mg/m2), once in the morning and once in the evening, taken orally within 30 minutes after meals. It is administered continuously for 14 days from day 1 to day 14, with a 21 day treatment cycle.
  Arms: Utidelone Capsule combination with Capecitabine
Drug: Utidelone Capsule (Part 3) — Utidelone capsule: 60 mg/m2/d, administered once a day on an empty stomach, continuously for 5 days from day 1 to day 5, with a treatment cycle of 21 days.
  Arms: Utidelone Capsule combination with Capecitabine

SUMMARY:
This study has three parts. Part 1 is a dose-escalation trial, Part 2 is a pharmacokinetic comparison and food effect study, and Part 3 is extended trial of combination of utidelone capsule and capecitabine. The primary objectives are 1. To evaluate the safety and tolerability of utidelone capsules in patients with advanced solid tumors and to determine the Maximum Tolerated Dose (MTD) and Dose Limiting Toxicity (DLT). 2. To evaluate the objective response rate in patients with advanced metastatic breast cancer treated with the combination of utidelone capsule and capecitabine. The secondary objectives are: 1. to evaluate the absolute bioavailability of utidelone capsules relative to utidelone injection; 2. to evaluate the pharmacokinetic profile of utidelone capsules in patients with advanced solid tumors; 3. to preliminarily evaluate the efficacy and safety of utidelone capsules in patients with advanced solid tumors; and 4. to recommend doses and dosing regimens for subsequent clinical trials. 5. To evaluate the Progression-Free Survival (PFS), safety and pharmacokinetics of utidelone capsule combined with capecitabine in the treatment of patients with advanced metastatic breast cancer.

DETAILED DESCRIPTION:
Part 1 is a dose-escalation trial, and it's an open design; Part 2 is a pharmacokinetic comparison and food effect study, and it's an open, controlled study;Part 3: Extended trial of combination of utidelone capsule and capecitabine.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled into the study:

1. Patients who have fully understood the objectives, content, process of the study and possible adverse events, voluntarily serves as a subject and signs the informed consent form.
2. Part 1 and Part 2: Patients with definitive histopathological diagnosis of advanced solid tumors. Part 3: Patients were diagnosed with advanced metastatic breast cancer by pathology and/or cytology.
3. Part 1 and Part 2: Male or female subjects aged ≥18 and ≤65, Part 3: Male or female subjects aged ≥18 and ≤70, with ECOG performance status scored 0-1.
4. Expected survival time ≥ 12 weeks;
5. At least one measurable lesion present according to RECIST 1.1 criteria.
6. Baseline routine blood tests within 1 week prior to enrollment is normal (not received blood transfusions or hematopoietic-stimulating factors within 14 days), with CTCAE grade ≤1 (based on normal values at each site's laboratory): a) Neutrophil count (ANC) ≥ 1.5 × 109/L; b) platelet count (PLT ) ≥ 100 × 109/L; c) Hemoglobin ≥9.0 g/dL.
7. Liver and kidney function test results are normal within 1 week prior to enrollment, with CTCAE grade ≤1 (based on normal values at each site's laboratory): a) Total bilirubin (TBIL) ≤ 1.5× the upper limit of normal value (ULN); b) Serum Glutamic Pyruvic Transaminase/Alanine Aminotransferease (SGPT /ALT) ≤ 2.5× ULN (Part 3 allowed ≤5×ULN in patients with liver metastases); c) Serum Glutamic-oxaloacetic Transaminase/Aspartate Aminotransferase (SGOT /AST) ≤ 2.5× ULN (Part 3 allowed ≤5×ULN in patients with liver metastases); d) Creatinine clearance (Ccr) ≥60 ml/min.
8. Patients with no functional disorders of major organs.
9. Fertile males and females of childbearing potential must agree to use effective contraception (so do their partners, using hormonal or barrier contraception, or abstinence) during the study and within at least 12 weeks after the last dose. The blood or urine pregnancy test for female patients of childbearing potential prior to enrollment must be negative.
10. Part 3: breast cancer patients who had received ≤4 previous chemotherapy regimens (adjuvant chemotherapy/neoadjuvant chemotherapy was considered as one chemotherapy regimen);
11. Part 3: history of prior treatment with at least one anthracycline or one taxane as neoadjuvant/adjuvant or advance therapy or both.

Exclusion Criteria:

Subjects who fulfill any one of the following exclusion criteria will be excluded from the study:

1. Patients who have received non-investigational anti-tumor therapies (such as chemotherapy, radiotherapy, immunotherapy, biological therapy or traditional Chinese medicine treatment) within 2 weeks prior to study drug administration.
2. Subjects with severe hypersensitivity to castor oil (this criteria is applicable to Part 2 of the study), and subjects who had hypersensitivity reaction caused by previous anti-microtubule drugs.
3. Patients with uncontrollable brain metastases (brain metastatic lesion confirmed by examination within 2 months after radiotherapy or other localized treatment); patients with uncontrollable bone metastases (patients who have had fracture or have the risk of fracture in recent days, patients who need surgery or localized radiotherapy in recent days, patients with other critical conditions)
4. Patients with serious comorbidities, such as severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infections, active peptic ulcers, etc.
5. Patients with mental illnesses which are hard to control, patients who lack legal capacity or have limited legal capacity.
6. Patients with gastrointestinal diseases such as esophageal obstruction, pyloric obstruction, intestinal obstruction, or who are post-operative of gastrointestinal resection, or who have difficulty in swallowing due to other factors, interfering with oral administration and absorption of the drug.
7. Patients with active hepatitis B infections.
8. Patients with peripheral neuropathy grade>1 within 4 weeks prior to enrollment (NCI CTCAE 5.0).
9. Patients who still experience ≥ Grade 2 acute toxicities caused by previous anti-tumor therapies (e.g. chemotherapy, radiotherapy, immunotherapy, biological therapy or TCM treatment) prior to enrollment (NCI-CTCAE 5.0, except alopecia).
10. Patients who have undergone any major surgery or have major trauma within 4 weeks prior to administration of the investigational product or are expected to undergo major surgery during the treatment.
11. Patients who have participated in another clinical trial or have received other investigational treatments within 4 weeks prior to administration of the investigational product.
12. Patients who, in the opinion of the investigator, are not suitable to participate in this study.
13. Part 3: other malignant tumors within 5 years before enrollment, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, thyroid papillary carcinoma;
14. Part 3: previous or current capecitabine therapy (except if capecitabine was used in neoadjuvant/adjuvant therapy and progression occurred > 12 months after completion of treatment, inclusion was allowed);
15. Part 3: patients with previous fluorouracil medication history with severe allergy or known dihydropyrimidine dehydrogenase (DPD) deficiency;
16. Part 3: previous or current use of utidelone (including utidelone injection and utidelone capsule); 17) Part 3: pregnant or lactating patients; 18) Part 3: uncontrolled pleural effusion, pericardial effusion or ascites (drainage once a month or more); 19) Part 3: a history of immunodeficiency, including positive HIV antibody test, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-03-09 (Estimated); Study Completion 2025-04-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose, MTD | 8 months
  The maximum tolerated dose (MTD) is defined as the highest dose tested in which none or only one patient experienced DLT attributable to the study drug(s), when 6 patients were treated at that dose and are evaluable for toxicity. The MTD is one dose level below the lowest dose tested in which 2 or more patients experienced DLT attributable to the study drug(s).
Dose-Limiting Toxicity, DLT | 8 months
  DLT is observed during Cycle 1 in the dose escalation trial. Any toxicity meeting the criteria outlined in the protocol, at least possibly related to study drug (i.e. definitely, probably, or possibly attributed), will be considered a DLT.
Objective Response Rate, ORR | 6 weeks
  To evaluate the objective response rate (ORR) of utidelone capsule combined with capecitabine in the treatment of patients with advanced metastatic breast cancer

SECONDARY OUTCOMES:
Bioavailability of Utidelone Capsule | 8 months
  Endpoint indicator: F
Maximum (or peak) serum concentration-Cmax | 8 months
  Cmax of Utidelone Capsule
Time to peak drug concentration-Tmax | 8 months
  Tmax of Utidelone Capsule
the area under the concentration-time curve from dosing (time 0) to time t-AUC0-t | 8 months
  the AUC0-t of Utidelone Capsule
the time required for plasma concentration of a drug to decrease by 50%-t1/2 | 8 months
  the t1/2 of Utidelone Capsule
Objective Response Rate-ORR | 12 months
  The percentage of patients who have a partial response or complete response to the treatment within a certain period of time.
Treatment-related Adverse Event-TRAE | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Progression-Free Survival, PFS | 6 weeks
  To evaluate the Progression-Free Survival (PFS) of eutidrone capsules combined with capecitabine in the treatment of patients with advanced metastatic breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No